CLINICAL TRIAL: NCT02138877
Title: Dismembered Pyeloplasty With and Without After Coming Stent in Neonatal Ureteropelvic Junction Obstruction
Brief Title: Dismembered Pyeloplasty With and Without After Coming Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohammed said elsheemy, Associte professor of urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61178
Record Dates: First submitted 2014-05-10; First posted 2014-05-15 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Pelviureteric Junction Obstruction; Pyeloplasty; Neonatal Hydronephrosis; Obstructive Uropathy; Urinary Stent
Keywords: Pelviureteric junction obstruction; pyeloplasty; Neonate affected by hydronephrosis; obstructive uropathy; urinary stent
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- After coming stent (Active Comparator): Dismembered pyeloplasty with insertion of an after coming stent
  Interventions: Procedure: After coming stent after dismembered pyeloplasty
- Stentless (Active Comparator): Stentless dismembered pyeloplasty
  Interventions: Procedure: Stentless dismembered pyeloplasty

INTERVENTIONS:
Procedure: After coming stent after dismembered pyeloplasty — Dismembered pyeloplasty through lumbar incision. The patients who are randomized to the after coming stent arm, an after coming stent is inserted. Distal part of it is positioned in the mid ureter. The proximal end is passed through the renal parenchyma (usually the lower kidney calyx) to be exteriorized through stab wound and fixed to the skin. The size of external stent is 4-5 F.
  Arms: After coming stent
Procedure: Stentless dismembered pyeloplasty — Dismembered pyeloplasty through lumbar incision. No stents are inserted
  Arms: Stentless

SUMMARY:
to compare outcome of pyeloplasty in pediatric population less than 6 months in age using an after coming stent versus stentless pyeloplasty.

DETAILED DESCRIPTION:
A prospective randomized control study including patients divided into two groups,all patient undergoes dismembered pyeloplasty First group will be with an after coming stent ,Second group will be stentless to compare outcome of pyeloplasty in pediatric population less than 6 months in age

ELIGIBILITY:
Inclusion Criteria:

* Pelvi-ureteric junction obstruction (PUJO)
* Asymptomatic obstruction with reduced function (less than 35-40%)
* Asymptomatic obstruction with antero-posterior diameter exceed 40 mm
* Asymptomatic obstruction with deterioration on conservative follow up.
* Symptomatic PUJ obstruction, e.g. pain, renal mass, fever and stones.

Exclusion Criteria:

* Secondary Pelvi-ureteric junction obstruction
* Solitary kidney
* Gross pyuria
* Ectopic kidney
* Dilated ureter

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Postoperative Hospital stay | 1 week
  Postoperative Hospital stay
Leakage | 1 week
  occurrence of post operative leakage
2ry intervention | 1 month
  Need for 2ry intervention in the form of insertion of ureteral stent
Fever | 1 month
  Postoperative fever

SECONDARY OUTCOMES:
Assessment of kidney function after repair | 6 months
  - Assessment of kidney function after repair using renogram and ultrasound
success | 6 months
  Need for 2ry treatment of persistent pelviureteric junction obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S ElSheemy, A professor, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt